CLINICAL TRIAL: NCT00087464
Title: Tenofovir, Emtricitabine, and Nevirapine for Recently HIV-Infected Subjects: Can Short-Course, Once Daily Therapy Reduce the Viral Load at 12 Months From Estimated Date of Infection?
Brief Title: Three Month Course of Anti-HIV Medications for People Recently Infected With HIV
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study was withdrawn before any participants were recruited and enrolled
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI-08-005; 11534 (Registry Identifier: DAIDS ES); AIEDRP AI-08-005
Record Dates: First submitted 2004-07-08; First posted 2004-07-13 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Acute Infection; Treatment Naive; Treatment Interruption
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine; Nevirapine; Tenofovir

INTERVENTIONS:
Drug: Emtricitabine
Drug: Nevirapine
Drug: Tenofovir disoproxil fumarate

SUMMARY:
Short-term therapy may reduce the amount of HIV in the blood of adults recently infected with HIV. The purpose of this study is to see whether it is better for people to take a short course of anti-HIV drugs when they are first infected or if it is better to wait until the HIV infection causes health problems before taking anti-HIV drugs.

DETAILED DESCRIPTION:
Limited access to HIV treatment is a major problem in many parts of the world. If a well tolerated anti-HIV regimen with convenient once-daily dosing is effective in reducing viral load in people with recent or early HIV infection, this regimen could be used globally for controlling HIV. This study will determine the effectiveness of a three-month antiretroviral regimen in reducing viral load in HIV infected adults who were recently infected or have recently seroconverted. This study will recruit participants from Alabama and Tennessee in the United States and in Lusaka, Zambia.

Participants in this study must also be enrolled in the AIEDRP CORE01 study. Participants in this study will be divided into Early and Acute groups. Participants in the Early group will be people who have recently seroconverted; participants in the Acute group will be people with primary HIV infection. All participants will choose to receive the once-daily dosing regimen of emtricitabine, nevirapine, and tenofovir disoproxil fumarate. Didanosine, efavirenz, and stavudine may be substituted for other drugs in the regimen at the investigator's discretion. Participants will take the three-drug regimen for 90 days. If a participant's CD4 count is higher than 350 cells/mm3 at Day 90, the participant will stop therapy. If a participant's CD4 count is 350 cells/mm3 or lower at Day 90, or if the participant's CD4 count drops to 350 cells/mm3 or lower while therapy is stopped, the participant will receive an additional 30 days of therapy. This therapy strategy may be repeated as necessary up to Day 180. All participants taking the three-drug regimen will be followed, regardless of whether or not they have taken the regimen beyond Day 90.

In addition to AIEDRP CORE01's study visits, 7 additional study visits will occur at pretreatment, on Day 3, and at Weeks 1, 3, 8, 16, and 20. Blood collection will occur at all study visits. Data from study participants will be compared with data from a historical cohort of previously identified HIV infected adults with acute or early infection who did not receive treatment but were followed prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Acute or early HIV infection, as determined by the NIH Acute Infection and Early Disease Research Program (AIEDRP) definition
* Coenrolled in AIEDRP CORE01 trial
* Willing to use acceptable methods of contraception

Exclusion Criteria:

* Any severe medical illness that, in the opinion of the investigator, will interfere with the ability to adhere to therapy or will result in making therapy too risky for the patient
* Significant psychiatric illness or ongoing substance abuse that, in the opinion of the investigator, will compromise the ability of the patient to follow study procedures safely and consistently
* Hepatitis B or C infection AND liver enzymes of Grade 2 or greater OR evidence or history of severe hepatitis or cirrhosis
* Creatinine clearance less than 50 ml/min
* Received more than one month of prior antiretroviral therapy. Women who received short-term dosing of nevirapine to prevent mother-to-child transmission during childbirth are not excluded if they meet other study requirements. They should only be given nevirapine as part of an initial study regimen if resistance testing can be done to confirm that they do not have nevirapine resistance.
* Coenrolled in any other HIV treatment or investigational drug trial
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Michael Kilby, MD, Principal Investigator — University of Alabama at Birmingham

REFERENCES:
- [Background] Babiker A, Darbyshire J, Pezzotti P, Porter K, Prins M, Sabin C, Walker AS; CASCADE Collaboration. Short-term CD4 cell response after highly active antiretroviral therapy initiated at different times from seroconversion in 1,500 seroconverters. J Acquir Immune Defic Syndr. 2003 Mar 1;32(3):303-10. doi: 10.1097/00126334-200303010-00010. PMID 12626891
- [Background] van Leth F, Phanuphak P, Ruxrungtham K, Baraldi E, Miller S, Gazzard B, Cahn P, Lalloo UG, van der Westhuizen IP, Malan DR, Johnson MA, Santos BR, Mulcahy F, Wood R, Levi GC, Reboredo G, Squires K, Cassetti I, Petit D, Raffi F, Katlama C, Murphy RL, Horban A, Dam JP, Hassink E, van Leeuwen R, Robinson P, Wit FW, Lange JM; 2NN Study team. Comparison of first-line antiretroviral therapy with regimens including nevirapine, efavirenz, or both drugs, plus stavudine and lamivudine: a randomised open-label trial, the 2NN Study. Lancet. 2004 Apr 17;363(9417):1253-63. doi: 10.1016/S0140-6736(04)15997-7. PMID 15094269
- See also: Click here for more information about AIEDRP CORE01 — http://clinicaltrials.gov/ct/show/NCT00086372